CLINICAL TRIAL: NCT03918863
Title: Effects of a Neuromuscular Electrical Stimulation Protocol in Women With Patellofemoral Pain
Brief Title: Neuromuscular Electrical Stimulation on Patellofemoral Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Jamilson Simões Brasileiro, Professor, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAM2019
Record Dates: First submitted 2019-04-02; First posted 2019-04-18 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-05

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: electromyography; physiotherapy; knee; quadriceps muscle
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular electrical stimulation (Experimental): 8-week exercise program, twice a week, with neuromuscular eletrical stimulation on vastus medialis and gluteus medius.
  Interventions: Other: Neuromuscular electrical stimulation
- Exercise (Active Comparator): 8-week exercise program, twice a week.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Neuromuscular electrical stimulation — Exercise protocol associated with neuromuscular electrical stimulation on vastus medialis and gluteus medius. Parameters: rectangular pulse shape, biphasic, symmetrical, pulse duration of 200μs, interbust interval of 10ms and frequency of 2.500Hz modulated in 50 bursts.
  Other Names: Muscular eletrical stimulation
  Arms: Neuromuscular electrical stimulation
Other: Exercise — Same protocol of exercises of the other group, without association of electrical stimulation.
  Arms: Exercise

SUMMARY:
Objective this study is to analyze the effects of an intervention protocol with neuromuscular electrical stimulation in the vastus medialis obliquus and gluteus medius (GM) associated with exercises on electromyographic activity, muscle performance, self-reported functionality and pain of women with patellofemoral pain.

DETAILED DESCRIPTION:
This is a randomized, blinded trial in which 40 women, aged 18-30 years, will be randomized into 2 groups: Stimulation and Exercise Group (SEG) - will perform an exercise protocol associated with stimulation in the vastus medialis (VM) and gluteus medius (GM) muscles. Exercises Group (ExG) - will perform the same protocol of exercises of the previous group, however, without association with neuromuscular electrical stimulation. The intervention will occur twice a week for eight weeks. All volunteers will be submitted to the evaluation of the electromyographic activity of the VM, the GM and the vastus lateralis, the dynamometric parameters, the intensity of the pain and the functionality, in four moments: 72h hours before the beginning of the intervention; after 4 weeks of intervention; after 8 weeks of intervention; after 16 weeks from the start of the intervention (eight weeks after the end of the protocol). In this way, the investigators will investigate the applicability of the proposed trial with the use of neuromuscular electrical stimulation and identify the effects of this resource in the treatment of PFP.

ELIGIBILITY:
Inclusion Criteria:

* Present anterior or retropatellar pain during at least two of the following functional activities: sitting for long periods, going up or down stairs, running, kneeling down, crouching or jumping;
* A minimum pain score of three on the numerical pain scale, at the last 24 hours, with insidious and non-traumatic onset of symptoms for at least one month.

Exclusion Criteria:

* History of surgery, trauma or an osteomioarticular system injury in the lower limbs in the last six months;
* Other pathology associated with the knee joint and could not have performed physical therapy treatment in the last twelve weeks;
* Body mass index greater than 30;
* Pregnancy or breastfeeding;
* Contraindications for the application of neuromuscular electrical stimulation;
* Intolerance or non-acceptance of electric current;
* Missing more than two intervention sessions.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Knee pain | Change from baseline in knee pain at 8 weeks.
  Evaluation of pain level in the knee using the Numerical Pain Scale, graded from 0 to 10, where 0 indicates absence of pain and 10 indicates the worst pain imaginable.
Knee function | Change from baseline in knee function at 8 weeks.
  Evaluation of knee function using the Anterior Knee Pain Scale, that is a questionnaire encompassing 13 items related to different levels of knee function, with scores ranging from zero (representing the highest possible deficit) to 100 (meaning that the subject does not present any deficit).

SECONDARY OUTCOMES:
Root Mean Square (RMS) | Change from baseline in RMS at 8 weeks.
  Evaluation of the amplitude oh the electromyographic sinal (RMS) of vastus medialis, vastus lateralis and gluteus medius.
Time of muscle activation (Onset) | Change from baseline in onset of the electromyographic at 8 weeks.
  Evaluation of time of muscle activation electromyographic (onset) of vastus medialis, vastus lateralis and gluteus medius.
Isokinetic performance | Change from baseline in peak torque normalized for body weight at 8 weeks.
  Evaluation of isokinetic variable peak torque normalized for body weight (%) of knee extensors and hip abductors.
Isokinetic performance | Change from baseline in average peak torque at 8 weeks.
  Evaluation of isokinetic variable average peak torque (Nm) of knee extensors and hip abductors.
Isokinetic performance | Change from baseline in average power at 8 weeks.
  Evaluation of isokinetic variable average power (W) of knee extensors and hip abductors.
Isokinetic performance | Change from baseline in total work at 8 weeks.
  Evaluation of isokinetic variable total work (J) of knee extensors and hip abductors.

CONTACTS AND LOCATIONS:
Overall Officials: Jamilson S Brasileiro, PhD, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (2):
- Brazil (2):
  - Universidade Federal do Rio Grande do Norte, Natal, Rio Grande do Norte
  - Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Melo SA, Macedo LB, Bullhoes LCC, Cavalcanti RL, Azevedo Rodolfo JI, Brasileiro JS. Effects of neuromuscular electrical stimulation on patellofemoral pain: A randomized controlled trial. J Bodyw Mov Ther. 2024 Jul;39:390-397. doi: 10.1016/j.jbmt.2024.03.022. Epub 2024 Mar 19. PMID 38876657